CLINICAL TRIAL: NCT01913067
Title: A Phase II Evaluating Cabazitaxel in Patients With Brain Metastasis Secondary to Breast and Non-small Cell Lung Cancer
Brief Title: Evaluation of Cabazitaxel in Patients With Brain Metastasis Secondary to Breast Cancer and NSCLC
Acronym: CRANIAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Scientific rationale is deemed obsolete. Funders lost interest in the trial.
Sponsor: Jules Bordet Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE2100; 2012-005194-32 (EudraCT Number)
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Brain Metastasis; Breast Cancer; Non Small Cell Lung Cancer
Keywords: brain metastasis; breast cancer; HER2 negative; NSCLC
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Eligible patients will receive intravenous 25mg/m2 cabazitaxel every 3 weeks. Contrast-enhanced whole brain MRI will be performed every two cycles. Patients who show ≥50% volumetric reduction in the size of the brain lesion(s) will continue on cabazitaxel until disease progression or unacceptable toxicity. Patients who show evidence of disease progression and/or developed progressive neurological symptoms will be taken off study and offered whole brain irradiation. Patients who do not meet both criteria can have the choice either to continue on study drug or to be taken off study according to the investigator discretion.
  Interventions: Drug: Cabazitaxel; Procedure: Contrast-enhanced whole brain MRI

INTERVENTIONS:
Drug: Cabazitaxel — Intravenous, 25 mg/m2 every 3 weeks
  Other Names: Jevtana
Procedure: Contrast-enhanced whole brain MRI — Evaluation of the volumetric reduction in the size of the brain lesion(s).

SUMMARY:
A phase II trial evaluating Cabazitaxel in patients with brain metastasis secondary to breast and non-small-cell lung cancer (NSCLC).

OBJECTIVES:

Primary:

The purpose of this study is to determine if cabazitaxel can induce a reduction in the size brain metastasis in metastatic HER2-negative breast cancer and NSCLC with brain metastasis who were not previously treated with whole brain irradiation or require immediate brain irradiation.

Secondary:

* To determine the effect of cabazitaxel on the time to initiating whole brain irradiation or radiosurgery
* To determine the effect of cabazitaxel on the time to developing neurological symptoms
* To determine the effect of cabazitaxel on the time to disease progression in the brain
* To determine the effect of cabazitaxel on the time to disease progression outside the brain. This will be evaluated separately for the breast and NSCLC cohorts To determine the objective extra-cranial response (if applicable). This will be evaluated separately in the breast and NSCLC cohorts
* To determine the safety of cabazitaxel

DETAILED DESCRIPTION:
This is a single arm, prospective trial using a 2-stage Simon design, in which eligible patients will receive intravenous cabazitaxel for two cycles followed by response evaluation. Based on the pre-specified criteria of response (intra-cranial, patient will be allowed to continue on study drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age>18, ECOG 0-1
* Histologically confirmed 1) HER2-negative invasive breast carcinoma or 2) NSCLC
* In patients with breast cancer, HER2-negative status by FISH or immunohistochemistry (score 0, or +1).
* In patients with breast cancer, known estrogen and progesterone receptor status.
* Evidence of measurable disease in the brain (at least 1cm)
* Stable or decreasing dosage of steroids for 7 days prior to baseline MRI.
* No evidence of (cortical) cognitive impairment as defined by a Mini-Mental Status Exam (MMSE) score ≥ 25/30.
* No more than 4 prior lines of systemic chemotherapy in the metastatic setting
* Adequate hematopoietic function defined as:

  * Hemoglobin ≥ 9.0g/dL
  * Absolute neutrophilic count ≥ 1.5 x 109L
  * Platelet count ≥ 100 x 109L
* Adequate hepatic function defined as:

  * AST ≤ 2.5 x upper limit of normal (ULN)
  * ALT ≤ 2.5 x ULN
  * Total bilirubin ≤ 1.0 x ULN
* Adequate renal function defined as serum creatinine ≤ 1.5 x ULN. If creatinine ranges from 1.0 - 1.5 x ULN, creatinine clearance determined by CKD-EPI formula should be calculated and only patients with clearance >60 mL/min are eligible
* Adequate contraceptive method in patients with child-bearing potential.

Exclusion Criteria:

* History of prior whole brain irradiation
* Progressive neurological symptoms requiring immediate brain irradiation
* Pregnancy or lactation
* History of hypersensitivity reaction to taxanes
* History of hypersensitivity to polysorbate 80 containing agents
* Current or planned treatment with strong inhibitors or inducers of cytochrome P450.
* Less than 3 weeks since the last treatment of chemotherapy, biological therapy, and/or immunotherapy
* Leptomeningeal carcinomatosis
* Contra-indication to contrast-enhanced MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of brain lesions. | week 6
  Objective response defined as a >= 50% volumetric reduction of brain lesions in the absence of increasing steroid use and progressive neurologic symptoms.

SECONDARY OUTCOMES:
Time to whole brain irradiation or radiosurgery | every 6 weeks until disease progression.
  Determine the effect of cabazitaxel on the time to initiating whole brain irradiation or radiosurgery
Time to developing neurological symptoms. | every 6 weeks until disease progression.
  Determine the effect of cabazitaxel on the time to developing neurological symptoms
Time to progression in the brain | every 6 weeks until disease progression.
  Determine the effect of cabazitaxel on the time to disease progression in the brain.
Time to progression extra-cranial | every 6 weeks until disease progression.
  Determine the effect of cabazitaxel on the time to disease progression outside the brain
Toxicity | every 3 weeks until 30 days after last treatment administration.
  Determine the safety of cabazitaxel

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, MD, PhD, Principal Investigator — Institute Jules Bordet
Locations (1):
- Institut Jules Bordet, Brussels, Brussels Capital, Belgium